CLINICAL TRIAL: NCT02569073
Title: Investigation of Cannabinoid Receptor Agonist Dronabinol in Patients With Functional Chest Pain
Acronym: ICAMP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22894
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Diseases
Keywords: Functional Chest Pain; Non-Cardiac Chest Pain; Esophageal Hypersensitivity
MeSH Terms: conditions — Esophageal Diseases | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dronabinol (Experimental): Patients who receive Dronabinol 5 mg, every other night, orally.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Patients who receive Placebo every other night, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol 5 mg, every other night, orally
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — Placebo--no drug
  Arms: Placebo

SUMMARY:
In a recent study, Dronabinol was shown to reduce symptoms in patients with Functional Chest Pain (non-cardiac chest pain). Additionally, metabolic measures and patients' weights were not adversely affected by this regiment. In fact, some cholesterol measures trended in a favorable direction with Dronabinol. The study lasted 28 days and patients took Dronabinol twice daily. The goal of this current study focuses on reducing the dose of Dronabinol to see if the same goals can be achieved. More so, the study will be extended to 12 weeks to gain a more longitudinal picture of therapy with Dronabinol. It is hypothesized that reducing the dose and extending the duration will continue to show an improvement in symptoms as well as no adverse metabolic outcomes.

DETAILED DESCRIPTION:
About 200,000 new cases of Functional Chest Pain (FCP) are diagnosed annually in USA. FCP is associated with poor quality of life and high health care expenditure. Gastroesophageal reflux disease (GERD), esophageal motility disorders, and psychological disorders may cause FCP. However, the mechanism(s) for FCP continue to be explored and include central and peripheral hypersensitivity as well as biomechanical dysfunction of the esophageal wall. CB1 receptor activation in synaptic clefts fine tunes neuronal firing and may in fact quell the over excitation associated with hypersensitivity.

Dronabinol, a cannabinoid receptor agonist with a preference for CB1 over CB2, is believed to reduce the esophageal hypersensitivity. CB1 receptors are located primarily on central and peripheral neurons (including the enteric nervous system) and myenteric plexus where they modulate neurotransmitter release. Activation of pre-junctional CB1 receptors may reduce excitatory enteric transmission and conceivably improve esophageal hyperreactivity and hypersensitivity, the hallmarks of FCP.

Previously, it was shown that Chest Pain Symptoms were greatly reduced when patients took 5 mg Dronabinol twice daily. Patients had very few side effects from this regiment although sedation was reported. The goal of this study focuses on reducing the dose of Dronabinol to 5 mg every other day, or essentially, one quarter of the dose. The effect of Dronabinol varies with CB1 receptor density in various tissues. It is hypothesized that at this reduced dose relief of chest pain will still be achieved without the sedating effects.

More so, Dronabinol at 5 mg twice daily failed to produce any adverse metabolic outcomes including measures of glucose, LDL, triglycerides, leptin, or transaminases. Dronabinol treatment tended to improve some of these measures although the study only lasted 28 days. Currently the hypothesis is that lower doses at a protracted time course will again fail to perturb homeostasis.

ELIGIBILITY:
Inclusion Criteria:

At least one episode of chest pain a week in the past month. Previous negative cardiac evaluation (EKG ± non invasive stress test ± coronary angiogram). Negative esophageal evaluation for a motility disorder (eg: achalasia) and GERD (normal endoscopy, normal 24 hr pH study, or unresponsive to 6 weeks of BID PPI therapy)

Exclusion Criteria:

1. Subjects requiring narcotics or other pain medications,
2. Subjects with known GERD (unless responsive to PPI therapy and on a stable dose), esophagitis, Barrett's esophagus or peptic stricture on endoscopy
3. Subjects with previous upper gastrointestinal surgery
4. Pregnancy
5. Subjects with diabetes, neuromuscular disorders, cardiac disorders, or other severe co-morbidities (Cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic).
6. Subjects with upper airway symptoms (such as hoarseness, wheezing or laryngospasm)
7. Medications such as baclofen, sucralfate and prokinetic agents or any agent considered a sedative, hypnotic, or psychoactive drug.
8. Known history of substance abuse.
9. Subject unable to consent.
10. Patient has history of comorbid psychiatric conditions including mania and schizophrenia. Patients will also be excluded who currently have a diagnosis of depression or undergoing treatment for depression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Chest Pain | Daily assessment for 12 weeks
  Patient will fill out a Chest Pain Questionnaire and symptom diary daily of symptoms which will be normalized to a numerical value for comparison among groups.

SECONDARY OUTCOMES:
Chest Pain Intensity | Daily assessment for 12 weeks
  Patient will fill out a Chest Pain Questionnaire and symptom diary daily of symptoms which will be normalized to a numerical value for comparison among groups.
GERD Symptom Checklist | Baseline, 2, 4, 8, and 12 weeks
  Patients will fill out a questionnaire pertaining to GERD symptoms which will be normalized to a numerical value for comparison among groups.
Short Form 36 | Baseline, 2, 4, 8, and 12 weeks
  A general health-related quality of life questionnaire that examines 8 domains: Physical Functioning, Role Functioning Physical, Role Functioning Emotional, Mental Health, Vitality, Bodily Pain, General Health, and Social Functioning
Esophageal Hypersensitivity and Distention | Baseline, 4, 8, and 12 weeks
  Sensory thresholds for first sensation, discomfort, and pain in the esophagus. Frequency, amplitude, area under the curve (AUC) of reactive esophageal contractions
Beck Depression Index | Baseline, 2, 4, 8, and 12 weeks
  Analysis of depressive symptoms normalized to a numerical value for comparison among groups.
Metabolic Parameters | Baseline, 2, 4, 8, and 12 weeks
  Total cholesterol will be measured and reported in mg/dL.
Weight | Baseline, 2, 4, 8, and 12 weeks
  Patient mass will be measured in kg.
Beck Anxiety Index | Baseline, 2, 4, 8, and 12 weeks
  Analysis of anxious symptoms normalized to a numerical value for comparison among groups.
Waist Circumference | Baseline, 2, 4, 8, and 12 weeks
  Patient's waist in cm will be measured.
Non-HDL Cholesterol | Baseline, 2, 4, 8, and 12 weeks
  Non-HDL cholesterol will be measured and reported in mg/dL.
HDL Cholesterol | Baseline, 2, 4, 8, and 12 weeks
  HDL cholesterol will be measured and reported in mg/dL.
Triglycerides | Baseline, 2, 4, 8, and 12 weeks
  Triglycerides will be measured and reported in mg/dL.
Glucose | Baseline, 2, 4, 8, and 12 weeks
  Glucose will be measured and reported in mg/dL.
Insulin | Baseline, 2, 4, 8, and 12 weeks
  Insulin will be measured and reported in µU/mL.
Leptin | Baseline, 2, 4, 8, and 12 weeks
  Leptin will be measured and reported in ng/mL.
ALT | Baseline, 2, 4, 8, and 12 weeks
  Leptin will be measured and reported in IU/L.
AST | Baseline, 2, 4, 8, and 12 weeks
  Leptin will be measured and reported in IU/L.
LDH | Baseline, 2, 4, 8, and 12 weeks
  LDH will be measured and reported in IU/L.
CRP | Baseline, 2, 4, 8, and 12 weeks
  CRP will be measured and reported in mg/L.

CONTACTS AND LOCATIONS:
Overall Officials: Ron W Schey, M.D., Principal Investigator — Temple University; Zachary W Reichenbach, M.D., Ph.D., Principal Investigator — Temple University; Henry Parkman, M.D., Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No